CLINICAL TRIAL: NCT03610269
Title: Spot-Check Noninvasive Hemoglobin (SpHb) Clinical Validation of INVSENSOR00026
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TORR0003
Record Dates: First submitted 2018-07-26; First posted 2018-08-01 (Actual); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- INVSENSOR00026 (Experimental): All enrolled subjects receive INVSENSOR00026 Pulse CO-Oximeter and sensor for the noninvasive measurement of hemoglobin (SpHb).
  Interventions: Device: INVSENSOR00026 (Pulse CO-Oximeter and sensor)

INTERVENTIONS:
Device: INVSENSOR00026 (Pulse CO-Oximeter and sensor) — Noninvasive Pulse CO-Oximeter and sensor that measures noninvasive hemoglobin (SpHb)

SUMMARY:
The primary objective of this clinical investigation is to evaluate the accuracy of using Masimo's INVSENSOR00026 Pulse CO-Oximeter and Sensor to measure hemoglobin, as compared to hemoglobin measurements obtained from various lab analyzer(s) and point of care device(s).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Subject has given written informed consent to participate in the study

Exclusion Criteria:

* (*) Pregnant or positive human chorionic gonadotropin (hCG) test
* (*) Any severe coagulopathy, chronic bleeding disorders (i.e., hemophilia) or recent thrombolysis
* (*) Hemoglobinopathies and synthesis disorders (i.e., sickle cell, thalassemias, etc.)
* (*) Subjects who are currently taking anticoagulant medication
* (*) Subjects with allergies to lidocaine, Pain Ease, latex, adhesives, or plastic
* (*) Subjects with skin abnormalities at the planned application sites that may interfere with sensor application, per directions-for-use (DFU) or trans-illumination of the site, such as psoriasis, eczema, angioma, burns, scar tissue, substantial skin breakdown, nail polish, acrylic nails, infections, abnormalities, etc.
* (*) Subjects unlikely to be able to refrain from excessive motion during data collection. Excessive motion includes postural changes, making hand gestures, involuntary muscular movements, etc.
* (*) Subjects with elevated blood pressure, skin or wrist abnormalities that may interfere with an arterial blood draw as determined by investigator or research medical staff.
* (*) Subjects who intend on participating in heavy lifting, repetitive movement of their wrist (including riding a motorcycle) or exercise (working out, riding a bike, etc.), or any activity that will put additional stress on the wrist within 24 hours following a study involving an arterial blood draw
* Subjects deemed not suitable for the study at the discretion of the investigator or research medical staff

Note: (*) May be self-reported by subject

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Torrance Clinical Research, Lomita, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INVSENSOR00026
Started | 143
Completed | 127
Not Completed | 16
Not completed — Physician Decision | 10
Not completed — Protocol Violation | 1
Not completed — Unable to draw blood | 1
Not completed — Screen fail | 4

BASELINE CHARACTERISTICS:
Population: Number of baseline participants excludes data from subjects with protocol deviations or those with insufficient blood sample volume.
Arm/Group | INVSENSOR00026
Number analyzed (Participants) | 111
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 101
  >=65 years | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 43
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 106
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 111

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Noninvasive Hemoglobin (SpHb) Measurement by Arms Calculation
Description: Accuracy of the INVSENSOR00026 will be determined by comparing the noninvasive hemoglobin measurement (SpHb) of the INVSENSOR00026 to the hemoglobin value obtained from a reference blood sample and calculating the accuracy root mean square (Arms) error value. In order to obtain the Arms value, the blood sample hemoglobin value is subtracted from the INVSENSOR00026 hemoglobin value for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: Up to 2 hours per subject
Measure: Number; unit: g/dL
Arm/Group | INVSENSOR00026
Number analyzed (Participants) | 111
g/dL | 0.93

ADVERSE EVENTS:
Time Frame: During the duration of the study and 2 weeks after participation in the study.
Arm/Group | INVSENSOR00026
All-Cause Mortality (participants affected / at risk) | 0/127
Serious Adverse Events (participants affected / at risk) | 0/127
Other Adverse Events (participants affected / at risk) | 2/127
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INVSENSOR00026 (N=127)
Vasovagal syncope (Injury, poisoning and procedural complications) | 1
Hematoma (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/69/NCT03610269/Prot_SAP_000.pdf